CLINICAL TRIAL: NCT05643976
Title: Assessing the Ability of KardioPAC, a Digital Tool, to Facilitate Lifestyle Change in Participants Enrolled in a Cardiac Rehabilitation Program
Brief Title: Investigating KardioPAC Mobile App to Improve Physical Fitness Among Cardiac Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: KURA Care (Unknown)
Responsible Party: Principal Investigator, Pam Taub, MD, Director of Step Family Foundation Cardiovascular Rehabilitation and Wellness Center Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 805399
Record Dates: First submitted 2022-11-16; First posted 2022-12-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Rehabilitation; Exercise; Quality of Life
MeSH Terms: conditions — Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-care cardiac rehabilitation (SOC CR) (Active Comparator)
  Interventions: Other: Standard of Care
- Cardiac Rehabilitation + KardioPAC (CR+KardioPAC) (Experimental)
  Interventions: Behavioral: KardioPAC Mobile Application; Other: Standard of Care

INTERVENTIONS:
Behavioral: KardioPAC Mobile Application — Like those in the SOC CR arm, participants assigned to the CR+KardioPAC arm will receive standard of care and attend CR as prescribed by their physician. Additionally, they will receive access to the digital app, KardioPAC, & a BP device for home use that will record their BP readings in the app.
  KardioPAC is a remote patient monitoring system that allows providers to monitor patients and send out daily reminders. It integrates with BP monitors and fitness watches to collect patient health information at home. The information is uploaded to the HIPAA-compliant server and presented on the website for providers to read. Its reminder system can be customized to meet diverse clinical needs.
  Lastly, the Kura Care in-house Registered Nurse will provide 20-30 min of health coaching to intervention arm participants on a weekly or bi-weekly basis via the app. The coaching will include greetings, review of medication adherence, encouragement to exercise, and symptom management, if applicable.
  Arms: Cardiac Rehabilitation + KardioPAC (CR+KardioPAC)
Other: Standard of Care — During the prescribed cardiac rehabilitation, the SOC CR intervention participants will receive standard of care by attending the 36-72 sessions of CR as prescribed by his/her physician and administered by the University of California San Diego Health Cardiac Rehabilitation Center.

SUMMARY:
The purpose of this study is to sustain regular physical activity, improve health-related quality of life, improve resting blood pressure, improve anthropometrics, and improve adherence to prescribed cardiac rehabilitation sessions among individuals referred for cardiac rehabilitation (CR). Numerous studies show that CR improves clinical outcomes in cardiovascular disease (CVD). Exercise as a reliable adjunctive intervention, however, remains limited due to poor short- and long-term adherence. This proposed study will examine the effectiveness of the Kura Care KardioPac digital application plus CR to significantly sustain exercise adherence among CR patients, as compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to the University of California San Diego Health Cardiac Rehabilitation Center for 36-72 sessions of intensive cardiac rehabilitation for one of the following medical conditions: myocardial infarction, coronary artery bypass surgery, stable angina, heart valve repair or replacement, coronary angioplasty or stenting, congestive heart failure, heart transplant, or peripheral arterial disease
2. Able to give informed consent in English
3. Able to perform study assessments as described
4. Resting BP<180/110 mmHg
5. Able to perform light to moderate exercise
6. Have not had a fall during the previous 6 months resulting in an injury
7. Clinical staff's permission to participate, including their assessment that participant is a good candidate for this research study
8. Ability to complete written or app-based surveys
9. Owns an Apple or Android mobile telephone capable of downloading and running the app

Exclusion Criteria:

1. Referred to CR following Ventricular Assist Device procedure
2. Angina not adequately managed with nitrates
3. Oxygen-dependent Chronic Obstructive Pulmonary Disease
4. Recent stroke or significant cerebral neurologic impairment that would interfere with participation.
5. Unable to operate a BP device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Delta change in minutes per week of moderate physical activity between baseline and end of study between SOC and intervention as measured by actigraphy. | ~4 Months
  Assess the ability of CR + KardioPAC as compared to standard-of-care CR to change the activity level of participants.

SECONDARY OUTCOMES:
Delta change in METs (Metabolic Equivalents of Task), a measure of the amount of oxygen consumed during activity compared to resting oxygen consumption. | ~4 Months
  Assess the ability of CR + KardioPAC as compared to standard-of-care CR to improve functional capacity (METs) at pre- and post-CR.

OTHER OUTCOMES:
Resting Blood Pressure | ~4 Months
  Assess the ability of CR + KardioPAC as compared to standard-of-care CR to change resting blood pressure at pre- and post-CR.
Body Composition | ~4 Months
  Assess the ability of CR + KardioPAC as compared to standard-of-care CR to change body composition at pre- and post-CR.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No